CLINICAL TRIAL: NCT00369707
Title: A Phase II Trial of Combination Bortezomib and Rituximab as Front-line Therapy for Low-grade Non-Hodgkin's Lymphoma
Brief Title: Trial of VELCADE and Rituxan as Front-line Tx for Low-grade NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 06H1; STU00005335 (Other: Northwestern University IRB)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2018-10

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib and Rituximab (Experimental): On days 1, 8, 15 and 22 of the 1st cycle, bortezomib will be administered intravenously (through a vein) over 3-5 seconds followed by an intravenous infusion of rituximab. How long it will take to infuse the dose of rituximab is dependent upon your weight and how well you tolerate the infusion; it is estimated this first infusion may take between 3-4 hours. During subsequent cycles, bortezomib will again be given on days 1, 8, 15 and 22. However, rituximab will only be given on day 1 of each cycle.
  Interventions: Drug: Rituximab; Drug: bortezomib

INTERVENTIONS:
Drug: Rituximab — On days 1, 8, 15 and 22 of the 1st cycle, bortezomib will be administered intravenously (through a vein) over 3-5 seconds followed by an intravenous infusion of rituximab. How long it will take to infuse the dose of rituximab is dependent upon your weight and how well you tolerate the infusion; it is estimated this first infusion may take between 3-4 hours. During subsequent cycles, bortezomib will again be given on days 1, 8, 15 and 22. However, rituximab will only be given on day 1 of each cycle.
  Other Names: Rituxan
Drug: bortezomib — On days 1, 8, 15 and 22 of the 1st cycle, bortezomib will be administered intravenously (through a vein) over 3-5 seconds followed by an intravenous infusion of rituximab. How long it will take to infuse the dose of rituximab is dependent upon your weight and how well you tolerate the infusion; it is estimated this first infusion may take between 3-4 hours. During subsequent cycles, bortezomib will again be given on days 1, 8, 15 and 22. However, rituximab will only be given on day 1 of each cycle.
  Other Names: Velcade, PS-341

SUMMARY:
Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with rituximab may kill more cancer cells.

This phase II trial is studying how well giving bortezomib together with rituximab works as first-line therapy in treating patients with low-grade B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a multicenter, prospective study.

* Induction therapy: Patients receive bortezomib IV over 3-5 seconds on days 1, 8, 15, and 22. Patients also receive rituximab IV on days 1, 8, 15, and 22 of course 1 and on day 1 of all subsequent courses. Treatment repeats every 35 days for 3 courses. Patients achieving a complete response, partial response, or stable disease proceed to maintenance therapy.
* Maintenance therapy: Beginning 6-8 weeks after induction therapy, patients receive bortezomib IV over 3-5 seconds and rituximab IV on day 1. Treatment repeats every 60 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples are collected at baseline and periodically during study treatment.

After completion of study therapy, patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed low-grade B-lymphocyte non-Hodgkins lymphoma
* Life expectancy > 12 months

Exclusion Criteria:

* No known history of HIV infection
* No other active infection
* No peripheral neuropathy ≥ grade 2 within the past 14 days
* No uncontrolled hypertension
* None of the following cardiac conditions:

  * Myocardial infarction within the past 6 months
  * No heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Electrocardiographic evidence of acute ischemia
  * Active conduction system abnormalities
* No serious medical or psychiatric illness that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior therapy for non-Hodgkins lymphoma
* No prior bortezomib or rituximab
* At least 3 weeks since prior chemotherapy, radiation therapy, immunotherapy, systemic anticancer biologic therapy, or anticancer hormonal therapy
* At least 2 weeks since prior investigational drugs
* No other concurrent systemic cytotoxic chemotherapy or investigational agents + No leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-08-09 (Actual); Primary Completion 2012-05-22 (Actual); Study Completion 2014-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M. Evens, DO, MS, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Evens AM, Smith MR, Lossos IS, Helenowski I, Millenson M, Winter JN, Rosen ST, Gordon LI. Frontline bortezomib and rituximab for the treatment of newly diagnosed high tumour burden indolent non-Hodgkin lymphoma: a multicentre phase II study. Br J Haematol. 2014 Aug;166(4):514-20. doi: 10.1111/bjh.12915. Epub 2014 Apr 25. PMID 24761968

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on August 8, 2006 with an accrual goal of up to 43 patients. The study was designed to enroll 15 patients initially to do an interim efficacy assessment. Accrual was suspended on November 14 2007 for this analysis and reopened on December 20, 2007. The study was closed on August 10, 2012 after 42 patients were enrolled.
Groups:
- Bortezomib and Rituximab: Induction Part A will be 1 cycle of 35 days. On days 1, 8, 15 and 22 of the cycle, bortezomib 1.6mg/m2 will be administered intravenously (through a vein) over 3-5 seconds followed by an intravenous infusion of rituximab 375mg/m2 which may take between 3-4 hours.
  Induction Part B will be up to 2 cycles of 35 days each. Bortezomib will be given on days 1, 8, 15 and 22. Rituximab will only be given on day 1 of each cycle.
  Maintenance period will be up to 4 cycles where 1 cycle= 2 months. Bortezomib and Rituximab will be given on day 1 of each cycle only.
Period: Induction Part A (1 Cycle -35 Days)
Arm/Group | Bortezomib and Rituximab
Started | 42
Completed | 42
Not Completed | 0
Period: Induction Part B (2 Cycles)
Arm/Group | Bortezomib and Rituximab
Started | 42
Completed | 35
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Not completed — Inadequate response/MD decision | 1
Not completed — Progressive disease | 1
Period: Maintenance Period (up to 4 Cycles)
Arm/Group | Bortezomib and Rituximab
Started | 35
Completed | 27
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — inadequate response/MD decision | 2
Not completed — Progressive disease | 4
Period: Follow up for 2 Years After Treatment
Arm/Group | Bortezomib and Rituximab
Started (All patients that receive treatment go into follow up at completion of study treatment.) | 41
Completed | 38
Not Completed | 3
Not completed — Death | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response and Partial Response) After Three Inductions Cycles of Treatment.
Description: The primary objective of this study is to assess the overall response rate. Overall response rate at this time point will be defined as complete response [CR] plus partial response [PR]) after 3 cycles of bortezomib/rituximab induction therapy for patients with previously untreated low-grade, B-cell NHL.
  Complete response requires complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities (e.g., lactate dehydrogenase [LDH]) definitely assignable to NHL. There must also be complete disappearance of lymphoma involvement in the bone marrow (if initially present).
  Partial response (PR) requires 50% decrease in SPD of the six largest dominant nodes or nodal masses and no increase in the size of the other nodes, liver, or spleen.
Time Frame: At baseline and at the completion of 3 cycles of treatment where 1 cycle equals 35 days.
Measure: Number; unit: percentage of patients
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
percentage of patients | 71

2. Secondary Outcome: Overall Response Rate After 1 Course of Induction Therapy
Description: Overall response rate (ORR) after 1 cycle of bortezomib/rituximab induction therapy.
  Overall response rate at this time point will be defined as complete response [CR] plus partial response [PR]) after 1 cycle of bortezomib/rituximab induction therapy for patients with previously untreated low-grade, B-cell NHL.
  Complete response requires complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities (e.g., lactate dehydrogenase [LDH]) definitely assignable to NHL. There must also be complete disappearance of lymphoma involvement in the bone marrow (if initially present).
  Partial response (PR) requires 50% decrease in SPD of the six largest dominant nodes or nodal masses and no increase in the size of the other nodes, liver, or spleen.
Time Frame: At baseline and at the completion of cycle 1 (1 cycle =35 days)
Measure: Number; unit: percentage of patients
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
percentage of patients | 33

3. Secondary Outcome: Overall Response Rate After Completion of Maintenance Therapy
Description: Overall response rate at completion of bortezomib/rituximab maintenance therapy.
  Overall response rate at this time point will be defined as complete response [CR] plus partial response [PR]) after 3 cycles of bortezomib/rituximab induction therapy and up to 4 cycles of maintenance for patients with previously untreated low-grade, B-cell NHL.
  Complete response requires complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities (e.g., lactate dehydrogenase [LDH]) definitely assignable to NHL. There must also be complete disappearance of lymphoma involvement in the bone marrow (if initially present).
  Partial response (PR) requires 50% decrease in SPD of the six largest dominant nodes or nodal masses and no increase in the size of the other nodes, liver, or spleen.
Time Frame: At baseline and every 2 months during treatment of up to 3 cycles of induction (1 cycle =35days) and 4 cycles of maintenance (1 cycle =2 months) for up to 12 months.
Measure: Number; unit: percentage of patients
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
percentage of patients | 71

4. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded)until the first date that recurrent or progressive disease is objectively documented.
  Complete response requires complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities (e.g., lactate dehydrogenase [LDH]) definitely assignable to NHL. There must also be complete disappearance of lymphoma involvement in the bone marrow (if initially present).
  Partial response (PR) requires 50% decrease in SPD of the six largest dominant nodes or nodal masses and no increase in the size of the other nodes, liver, or spleen.
  Progressive disease (PD) requires the appearance of any new lesion or increase by > 50% in the size of previously involved sites.
Time Frame: Every 2 months for up to 12 months then every 6 months for 2 years and annually for 1 year
Population: Data was not collected or analyzed for duration of response.
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Patients That Experience Adverse Events With Bortezomib/Rituximab Combination Treatment
Description: Assess the safety and tolerance of bortezomib/rituximab as induction and maintenance therapy. Data will be collected for grade 3 and grade 4 adverse events experienced by patients that are determined to be at least possibly related to at least one study drug. Toxicity data for bortezomib/rituximab will be collected on day 1 of every cycle (1 cycle = 35 days) for up to 7 cycles during treatment according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Day 1 of each cycle and at the completion of cycles 1 and 3, during treatment up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
Participants
  Neutropenia | 2
  Fever | 2
  Infection | 2
  Infusion reaction (rituximab) | 2
  Cardiac | 2
  Fatigue | 2
  Throbocytopenia | 1
  Diarrhea | 1
  Hypokalemia | 1
  Bowel obstruction | 1
  Dehydration | 1

6. Secondary Outcome: Tissue Evaluation
Description: Tissue microarray analysis from paraffin embedded tissue, gene expression profiling from frozen tissue (both from initial node biopsy collected/stored) and whole blood analysis of FCγR polymorphism
Time Frame: At baseline and at response assessment 1 after induction part A, 2, after induction part B and 3, maintenance period.
Population: Insufficient tumor samples were submitted for insufficient number of patients. No data was collected or analyzed.
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 0

7. Secondary Outcome: Correlation of Tumor Burden
Description: Correlation of tumor burden according to Groupe D'Etude des Lymphomes Follicularies (GELF) with recently developed Follicular Lymphoma International Prognostic Index (FLIPI) prognostic index. All patients enrolled in the study were required to have high tumor burden (HTB) as defined by GELF, where HTB is defined as representing higher risk disease and poorer outcomes than low tumor burden (LTB). Patients were put into low risk or high risk FLIPI groups. Low risk group with a score of 0-2 and high risk group with a score of 3-5.
  A FLIPI score of 0 to 1 = "low risk" with a 10 year overall survival of 70%. A score of 2= "intermediate risk" with a 10 year overall survival of 50%. Finally, a score of ≥ 3 is considered "high risk" with a 10 year overall survival of 35%. Data was collected in connection with high or low risk FLIPI and Progression Free Survival (PFS) or Overall Survival (OS) and is reported as percentage patient with high/low risk that are progression free or alive.
Time Frame: At the start of treatment and at Median follow up for all patients was 50 months (range 12-78 months) and on intent to treat, PFS and OS for all patients is reported at 4 years.
Measure: Number; unit: percentage of patients
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
percentage of patients
  4 year PFS high risk FLIPI | 26
  4 year PFS low risk FLIPI | 60
  4 year OS high risk FLIPI | 81
  4 year OS low risk FLIPI | 92

8. Secondary Outcome: Percentage of Patients With Treatment Failure
Description: Time to Treatment Failure (TTF) rate measured, from the time of first treatment to disease progression, relapse, second tumor, death from any cause, treatment toxicity requiring termination from the study, or for any reason treatment is discontinued permanently.
Time Frame: Median follow up for all patients was 50 months and on intent to treat, TTF rate for all patients is reported at 4 years.
Measure: Number; unit: percentage of patients
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
percentage of patients | 26

9. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: Progression Free Survival is measured from the time of first induction infusion to disease progression, relapse, second tumor, or death from any cause.
  Progressive disease (PD) requires the following:
  1. Appearance of any new lesion or increase by > 50% in the size of previously involved sites.
  2. Increase of > 50% in the SPD from nadir measurement of all involved dominant lymph nodes and liver nodules and spleen nodules or unequivocal progression in any non measurable disease or nondominant site.
  3. > 50% increase in greatest diameter of any previously identified node greater than 1 cm in its short axis or in the SPD of more than one node
Time Frame: Median follow up for all patients was 50 months (range 12-78 months) and on intent to treat, PFS for all patients is reported at 4 years.
Measure: Number; unit: percentage of patients
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
percentage of patients | 44

10. Post Hoc Outcome: Overall Survival Rate
Description: Overall survival (OS) will be measured from the time of first treatment to death from any cause.
Time Frame: Median follow up for all patients was 50 months (range 12-78 months) and on intent to treat, OS rate for all patients is reported at 4 years.
Measure: Number; unit: percentage of patients
Arm/Group | Bortezomib and Rituximab
Number analyzed (Participants) | 42
percentage of patients | 87

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the whole study over a 6 year and 4 month period. On average adverse event information for each patient was collected during patients treatment, for a maximum of 12 months.
Description: Adverse events were collected via systematic assessment during patients treatment visit days.
Arm/Group | Bortezomib and Rituximab
All-Cause Mortality (participants affected / at risk) | 6/42
Serious Adverse Events (participants affected / at risk) | 7/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Rituximab (N=42)
Diastolic heart failure (Cardiac disorders) | 1 (1)
Congestive Heart Failure exacerbation (Cardiac disorders) | 1 (1)
Anal squamous cell carcinoma (Congenital, familial and genetic disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Fever with normal ANC (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Lumbar disk pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fainting episode (Syncope) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Rituximab (N=42)
Allergic reaction/hypersensitivity (Immune system disorders) | 14 (16)
Allergic rhinitis (Immune system disorders) | 10 (10)
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 18 (28)
Neutrophils (neutropenia) (Blood and lymphatic system disorders) | 10 (15)
Leukocytes (total white blood cells) (Blood and lymphatic system disorders) | 19 (27)
Lymphopenia (Blood and lymphatic system disorders) | 24 (38)
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 14 (15)
Fatigue (General disorders) | 24 (24)
Fever (General disorders) | 8 (9)
Insomnia (General disorders) | 5 (5)
Rigors (General disorders) | 3 (3)
Sweating (General disorders) | 7 (8)
Weight loss (General disorders) | 7 (7)
Flushing (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 7 (7)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11 (13)
Anorexia (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 22 (29)
Abdominal distension/bloating (Gastrointestinal disorders) | 3 (3)
Mucositis/stomatitis (Gastrointestinal disorders) | 4 (4)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 25 (30)
Vomiting (Gastrointestinal disorders) | 10 (11)
Upper airway infection (Infections and infestations) | 3 (3)
Eye infection (Infections and infestations) | 4 (4)
Infection (NOS) (Infections and infestations) | 3 (3)
Edema (Blood and lymphatic system disorders) | 4 (4)
Edema in limbs (Blood and lymphatic system disorders) | 5 (6)
Transaminase (Metabolism and nutrition disorders) | 6 (6)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (4)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5 (5)
Albumin, serum low (Metabolism and nutrition disorders) | 5 (5)
Bilirubin, serum high (Metabolism and nutrition disorders) | 8 (8)
Bicarbonate- low (Metabolism and nutrition disorders) | 3 (3)
Creatinine, serum high (Metabolism and nutrition disorders) | 3 (5)
Calcium, serum low (Metabolism and nutrition disorders) | 5 (6)
Glucose, serum high (Metabolism and nutrition disorders) | 18 (24)
Glucose, serum low (Metabolism and nutrition disorders) | 6 (6)
Lactic acid dehydrogenase (LDH) (Metabolism and nutrition disorders) | 4 (9)
Magnesium, serum low (Metabolism and nutrition disorders) | 3 (3)
Potassium, serum high (Metabolism and nutrition disorders) | 4 (8)
Potassium, serum low (Metabolism and nutrition disorders) | 6 (10)
Sodium, serum high (Metabolism and nutrition disorders) | 3 (3)
Uric acid, serum high (Metabolism and nutrition disorders) | 3 (3)
Sensory neuropathy (Nervous system disorders) | 10 (11)
Pain in abdomen (Gastrointestinal disorders) | 5 (6)
Pain in extremity - limb (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in joints (Musculoskeletal and connective tissue disorders) | 4 (5)
Headache (Nervous system disorders) | 7 (7)
General pain NOS (General disorders) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Shortness of breath (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Swelling of the eye (Eye disorders) | 4 (5)
Flu like syndrome (General disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes